CLINICAL TRIAL: NCT00558272
Title: A Phase II, Randomised, Open-Label, Pilot Study to Evaluate the Safety and Effects on Bone Resorption of AZD0530 in Patients With Prostate Cancer or Breast Cancer With Metastatic Bone Disease.
Brief Title: Study to Evaluate the Safety and Effects AZD0530 on Prostate and Breast Cancer Subjects With Metastatic Bone Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8180C00034
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer; Prostate Cancer; Bone Neoplasms
Keywords: breast cancer; prostate cancer; metastatic bone disease; Subjects with breast cancer or prostate cancer with metastatic bone disease
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Bone Neoplasms; Bone Diseases | interventions — saracatinib; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZD0530 175 mg (Experimental): AZD0530 (saracatinib) 175 mg once daily
  Interventions: Drug: AZD0530
- Zoledronic Acid 4 mg (Experimental): Zoledronic Acid 4 mg on Day 1 of the 4-week treatment period
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: AZD0530 — Daily oral dose
  Other Names: Saracatinib
  Arms: AZD0530 175 mg
Drug: Zoledronic Acid
  Other Names: Zometa
  Arms: Zoledronic Acid 4 mg

SUMMARY:
The purpose of this study is to determine the effect of AZD0530 on subjects with breast cancer or prostate cancer with metastatic bone disease in comparison to zoledronic acid.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years or older with Prostate Cancer or Breast Cancer with Metastatic Bone Disease Have evidence of recurrence or disease progression
* At least one radiographically confirmed metastatic bone lesion
* No change of cancer therapy for at least 8 weeks before randomization

Exclusion Criteria:

* Have had any prior exposure to bisphosphonate
* Have had hip fractures or bilateral hip prothesis fracture of any kind or surgery to bone within the past 12 months
* Inadequate renal function or low haemoglobin
* Inadequate liver function as demonstrated by serum bilirubin ≥2 times the upper limits of reference range (ULRR) or by alanine aminotransferase (ALT), aspartate aminotransferase(AST) or ALP ≥2.5 times the ULRR (≥5 times the ULRR in the presence of liver metastases). If bone metastases are present and liver function is otherwise considered adequate by the investigator then elevated ALP will not exclude the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Finkelman, DDS, PhD, Study Director — AstraZeneca; Meabe Aklilu, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (28):
- United States (9):
  - Research Site, Pleasant Hill, California
  - Research Site, Sacramento, California
  - Research Site, Middlebury, Connecticut
  - Research Site, Aventura, Florida
  - Research Site, Baltimore, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Poughkeepsie, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Hershey, Pennsylvania
- Canada (5):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Denmark (4):
  - Research Site, Arhus N
  - Research Site, Frederica
  - Research Site, Herlev
  - Research Site, Holstebro
- Norway (2):
  - Research Site, Kristiansand
  - Research Site, Oslo
- Research Site, Lisbon, Portugal
- Spain (3):
  - Research Site, Barcelona, Catalonia
  - Research Site, Lleida, Catalonia
  - Research Site, Valencia, Valencia
- Research Site, Uppsala, Sweden
- United Kingdom (3):
  - Research Site, Cardiff
  - Research Site, Glasgow
  - Research Site, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomised=full analysis set: AZD0530 175mg=69, Zoledronic acid 4mg=70; safety set: AZD0530 175mg=68, Zoledronic acid 4mg=69
Period: Overall Study
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Started | 69 (Randomised) | 70 (Randomised)
30 Days Follow-up | 41 (30 days after last dose) | 67 (30 days after last dose)
Completed | 56 (4-week treatment period) | 68 (4-week treatment period)
Not Completed | 13 | 2
Not completed — Adverse Event | 10 | 0
Not completed — Death | 1 | 0
Not completed — Dev. of study specific discon. criteria | 1 | 0
Not completed — AZ study team decision | 0 | 1
Not completed — Incorrectly enrolled | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg | Total
Number analyzed (Participants) | 69 | 70 | 139
Age Continuous [Mean (Standard Deviation); unit: Years] | 67.6 (8.35) | 67.3 (11.58) | 67.4 (10.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 58 | 58 | 116

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Serum Beta C-terminal Cross-linking Telopeptide of Type I Collagen (betaCTX) at Week 4
Description: Result at Week 4 minus result at baseline as a percentage of the result at baseline, based on log transformed data. Back transformation of the least squares (LS) mean.
Time Frame: Baseline to Week 4
Population: The number of participants analyzed reflected the number of paired serum samples per participant that yielded valid assay results, not the total number of participants or completers. The number of evaluable paired serum samples will therefore be a subset of the total number of participants.
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage change in betaCTX
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 46 | 65
Percentage change in betaCTX | -71.1 [-75.9 to -65.4] | -68.4 [-73.0 to -63.2]

2. Secondary Outcome: Percentage Change From Baseline in Serum Bone-specific Alkaline Phosphatase (bALP) at Week 4
Description: as for outcome 1
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage change in bALP
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 48 | 66
Percentage change in bALP | -13.2 [-24.4 to -0.3] | -3.1 [-13.9 to 9.1]

3. Secondary Outcome: Percentage Change From Baseline in Serum Cross-linked C-terminal Telopeptide of Type I Collagen (ICTP) at Week 4
Description: as for outcome 1
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage change in ICTP
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 47 | 66
Percentage change in ICTP | -40.2 [-46.3 to -33.4] | 7.4 [-2.0 to 17.7]

4. Secondary Outcome: Percentage Change From Baseline in Serum N-terminal Propeptide of Type I Procollagen (PINP) at Week 4
Description: as for outcome 1
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage change in PINP
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 48 | 66
Percentage change in PINP | -26.1 [-36.0 to -14.7] | -29.5 [-37.7 to -20.3]

5. Secondary Outcome: Percentage Change From Baseline in Serum Tartrate-resistant Acid Phosphatase 5b (TRAP5b) at Week 4
Description: as for outcome 1
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage change in TRAP5b
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 48 | 65
Percentage change in TRAP5b | -36.9 [-42.7 to -30.4] | -43.4 [-48.0 to -38.4]

6. Secondary Outcome: Percentage Change From Baseline in Urine N-terminal Cross-linking Telopeptide of Type I Collagen Normalised to Creatinine (NTx/Cr) at Week 4
Description: as for outcome 1
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage change in NTx/Cr
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 46 | 62
Percentage change in NTx/Cr | -57.2 [-65.7 to -46.6] | -70.1 [-75.4 to -63.8]

7. Secondary Outcome: Percentage Change From Baseline in Urine Alpha-alpha C-terminal Cross-linking Telopeptide of Type I Collagen Normalised to Creatinine (aaCTx/Cr) at Week 4
Description: as for outcome 1
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage change in aaCTx/Cr
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 41 | 49
Percentage change in aaCTx/Cr | -68.2 [-76.7 to -56.5] | -82.8 [-87.1 to -77.0]

8. Secondary Outcome: Saracatinib: Area Under the Curve at Steady State (AUCss)
Description: Previous studies have shown that saracatinib reduces osteoclast function and bone resorption. Bone turnover, the combined result of bone formation and bone resorption, can be assessed in real time by measuring specific markers of bone turnover in serum and in urine. These markers were assessed in a study of patients with metastatic bone disease treated with saracatinib. Specific assays are available to quantitate these markers in serum and urine. In this study the effects of saracatinib on bone turnover were compared with the effects of zoledronic acid, a marketed drug known to inhibit bone resorption in cancer patients with bone metastatses.
Time Frame: Pre-dose on days 8, 15, 29; 2 hours, 4 hours, 6 hours, 9 hours post dose on day 29
Measure: Median (Full Range); unit: ng•hr/ml
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 51 | 0
ng•hr/ml | 7261 [3960 to 21500] |

9. Secondary Outcome: Saracatinib: Plasma Clearance at Steady State (CLss/F)
Time Frame: Pre-dose on days 8, 15, 29; 2 hours, 4 hours, 6 hours, 9 hours post dose on day 29
Measure: Median (Full Range); unit: L/h
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 51 | 0
L/h | 24.10 [8.15 to 44.2] |

10. Secondary Outcome: Saracatinib: Maximum Plasma Concentration at Steady State (Css,Max)
Time Frame: Pre-dose on days 8, 15, 29; 2 hours, 4 hours, 6 hours, 9 hours post dose on day 29
Measure: Median (Full Range); unit: ng/ml
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 51 | 0
ng/ml | 396.0 [190 to 1170] |

11. Secondary Outcome: Saracatinib: Minimum Plasma Concentration at Steady State (Css,Min)
Time Frame: Pre-dose on days 8, 15, 29; 2 hours, 4 hours, 6 hours, 9 hours post dose on day 29
Measure: Median (Full Range); unit: ng/ml
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 51 | 0
ng/ml | 229.0 [99.1 to 770] |

12. Secondary Outcome: Saracatinib: Time to Cssmax (Tmax)
Time Frame: Pre-dose on days 8, 15, 29; 2 hours, 4 hours, 6 hours, 9 hours post dose on day 29
Measure: Median (Full Range); unit: h
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 51 | 0
h | 4.0 [2 to 9] |

13. Secondary Outcome: N-desmethyl Metabolite of Saracatinib: Area Under the Curve at Steady State (AUCss)
Time Frame: Pre-dose on days 8, 15, 29; 2 hours, 4 hours, 6 hours, 9 hours post dose on day 29
Measure: Median (Full Range); unit: ng.h/ml
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 51 | 0
ng.h/ml | 1069 [529 to 5100] |

14. Secondary Outcome: N-desmethyl Metabolite of Saracatinib: Maximum Plasma Concentration at Steady State (Css,Max)
Time Frame: Pre-dose on days 8, 15, 29; 2 hours, 4 hours, 6 hours, 9 hours post dose on day 29
Measure: Median (Full Range); unit: ng/ml
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 51 | 0
ng/ml | 62.80 [25.3 to 253] |

15. Secondary Outcome: N-desmethyl Metabolite of Saracatinib: Minimum Plasma Concentration at Steady State (Css,Min)
Time Frame: Pre-dose on days 8, 15, 29; 2 hours, 4 hours, 6 hours, 9 hours post dose on day 29
Measure: Median (Full Range); unit: ng/ml
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 51 | 0
ng/ml | 34.30 [16.6 to 230] |

16. Secondary Outcome: N-desmethyl Metabolite of Saracatinib: AUCss Metabolite to Parent Ratio
Time Frame: Pre-dose on days 8, 15, 29; 2 hours, 4 hours, 6 hours, 9 hours post dose on day 29
Measure: Median (Full Range); unit: Ratio
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 51 | 0
Ratio | 0.1420 [0.081 to 0.354] |

17. Secondary Outcome: N-desmethyl Metabolite of Saracatinib: Time to Cssmax (Tmax)
Time Frame: Pre-dose on days 8, 15, 29; 2 hours, 4 hours, 6 hours, 9 hours post dose on day 29
Measure: Median (Full Range); unit: h
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 51 | 0
h | 2.0 [2 to 9] |

ADVERSE EVENTS:
Description: safety set: AZD0530 175mg=68, Zoledronic acid 4mg=69
Arm/Group | AZD0530 175 mg | Zoledronic Acid 4 mg
Serious Adverse Events (participants affected / at risk) | 11/68 | 4/69
Other Adverse Events (participants affected / at risk) | 51/68 | 46/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD0530 175 mg (N=68) | Zoledronic Acid 4 mg (N=69)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
General Physical Health Deterioration (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Viral Infection (Infections and infestations) | 1 | 0
Blood Creatinine Increased (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD0530 175 mg (N=68) | Zoledronic Acid 4 mg (N=69)
Nausea (Gastrointestinal disorders) | 16 | 3
Diarrhoea (Gastrointestinal disorders) | 13 | 4
Constipation (Gastrointestinal disorders) | 10 | 5
Vomiting (Gastrointestinal disorders) | 7 | 5
Influenza Like Illness (General disorders) | 3 | 8
Pyrexia (General disorders) | 4 | 6
Fatigue (General disorders) | 5 | 4
Asthenia (General disorders) | 4 | 1
Oedema Peripheral (General disorders) | 4 | 2
Influenza (Infections and infestations) | 0 | 11
Urinary Tract Infection (Infections and infestations) | 6 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 8 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 8 | 4
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Headache (Nervous system disorders) | 5 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2

LIMITATIONS AND CAVEATS:
Non-compliant patients were excluded from the biomarker analysis, in order to accurately assess effects due to treatment. The compliance criteria did not apply to the zoledronic acid arm, which led to an imbalance in the number of subjects analysed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a Study Site, or an investigator, requests permission to publish data from this study, any such publication (including oral presentations) is to be agreed with AstraZeneca prior to publication.